CLINICAL TRIAL: NCT01781572
Title: A Phase Ib/II, Multicenter, Open Label, Study of LEE011 in Combination With MEK162 in Adult Patients With NRAS Mutant Melanoma
Brief Title: A Phase Ib/II Study of LEE011 in Combination With MEK162 in Patients With NRAS Mutant Melanoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMEK162X2114; C4211005 (Other: Pfizer)
Record Dates: First submitted 2013-01-24; First posted 2013-02-01 (Estimated); Results first posted 2020-08-12 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-11

CONDITIONS: Locally Advanced or Metastatic NRAS Mutant Melanoma
MeSH Terms: interventions — ribociclib; binimetinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phase Ib (Experimental): The phase Ib is the dose escalation part where successive cohorts of 3-6 newly enrolled patients receiving various dose pairs considering the recommendation from an adaptive BLRM incorporating the EWOC principle until MTD(s)/RP2D is defined. If multiple alternate dosing schedules are explored in parallel, the allocation of patients will proceed in an alternating fashion. Approximately 40 patients are expected to be treated during the phase Ib part of the study.
  Dosing Schedule 1: MEK162 administered orally twice daily on a continuous dosing schedule. LEE011 administered orally once daily for 21 days followed by a 1 week break (28-day cycle).
  Dosing Schedule 2: MEK162 administered orally twice daily and LEE011 administered orally once daily for 3 weeks followed by a 1 week break (28-day cycle).
  Dosing Schedule 3: MEK162 administered orally twice daily and LEE011 administered once daily for 2 weeks followed by a 1 week break (21-day cycle).
  Interventions: Drug: LEE011; Drug: MEK162
- Phase II (Experimental): The Phase II part will begin once the MTD(s)/RP2D have been determined in the Phase Ib in order to assess antitumor activity of the LEE011and MEK162 combination. Patients enrolled in the Phase II part of the study are required to have measurable disease. Approximately 40 patients will be treated in this part.
  Phase II part will begin at the RP2D on the chosen schedule in order to assess antitumor activity of the LEE011 and MEK162 combination.
  Interventions: Drug: LEE011; Drug: MEK162

INTERVENTIONS:
Drug: LEE011 — LEE011 will be administered orally once daily
Drug: MEK162 — MEK162 will be administered orally twice daily

SUMMARY:
In the phase Ib, the primary purpose is to establish the maximum tolerated dose (MTD)(s)/recommended phase ll dose (RP2D) and schedule of LEE011 and MEK162 orally administered combination. Once the MTD(s)/RP2D have been determined for each tested schedule, additional patients will be enrolled in the phase II portion of the study at the RP2D on the chosen schedule in order to assess the anti-tumor activity of the combination in addition to continued evaluation of safety.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 1.
* Patients enrolled into phase Ib may be enrolled with evaluable disease only. Patients enrolled into the phase II expansion must have at least one measurable lesion as defined by RECIST 1.1 criteria for solid tumors.
* Patients must have adequate organ function, as defined by the following parameter

  1. Absolute Neutrophil Count (ANC) ≥ 1.5 x 109/L.
  2. Hemoglobin (Hgb) ≥ 9 g/dL.
  3. Platelets ≥ 75 x 109/L without transfusions within 21 days before 1st treatment.
  4. PT/INR and aPTT ≤ 1.5 ULN.
  5. Serum creatinine ≤1.5 ULN.
  6. Serum total bilirubin ≤ 1.5 x upper limit of normal (ULN).
  7. AST and ALT ≤ 3 x ULN, except in patients with tumor involvement of the liver who must have AST and ALT ≤ 5 x ULN.

Exclusion Criteria:

* Presence of any brain metastases detected by MRI or CT with i.v. contrast of the brain at screening.
* Uncontrolled arterial hypertension despite medical treatment
* Impaired cardiac function or clinically significant cardiac diseases, including any of the following:

  1. Left ventricular ejection fraction (LVEF) < 50% as determined by multiple gated acquisition scan (MUGA) or echocardiogram (ECHO).
  2. Congenital long QT syndrome or family history of unexpected sudden cardiac death.
  3. QTcF corrected with Frederica's or Bazett's formula QTcB >450 ms for males and >470 ms for females on screening ECG.
  4. Angina pectoris ≤ 3 months prior to starting study drug
  5. Acute myocardial infarction ≤ 3 months prior to starting study drug
  6. Clinically significant resting bradycardia
  7. History or presence of ventricular tachyarrhythmia
  8. Unstable atrial fibrillation (ventricular response >100 bpm)
  9. Complete left bundle branch block
  10. Right bundle branch block and left anterior hemi block (bifascicular block)
  11. Obligate use of a cardiac pacemaker or implantable cardioverter defibrillator
  12. Any other clinically significant heart disease
* Patients who are currently receiving treatment with agents that are known to cause QTc prolongation in humans.
* Patients who have neuromuscular disorders that are associated with elevated CK (e.g., inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy) or elevated baseline CK levels (≥ Grade 2)
* Patients who are currently receiving treatment with agents that are metabolized predominantly through CYP3A4 and that have a narrow therapeutic window.
* Patients with concurrent severe and/or uncontrolled concurrent medical conditions that could compromise participation in the study (i.e. uncontrolled diabetes mellitus, clinically significant pulmonary disease, clinically significant neurological disorder, active or uncontrolled infection).
* History or current evidence of retinal vein occlusion (RVO) or current risk factors for RVO (e.g. uncontrolled glaucoma or ocular hypertension, history of hyperviscosity or hypercoagulability syndromes).

Other protocol related inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2013-06; Primary Completion 2018-01-15 (Actual); Study Completion 2018-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (17):
- United States (7):
  - University of California, Dept of Oncology, San Francisco, California
  - California Pacific Medical Center Onc Dept, San Francisco, California
  - Karmanos Cancer Institute Dept of Oncology, Detroit, Michigan
  - Memorial Sloan Kettering Cancer Center Dept Oncology, New York, New York
  - Columbia University Medical Center- New York Presbyterian Onc Dept., New York, New York
  - Vanderbilt University Medical Center SC - Dept of Oncology ., Nashville, Tennessee
  - University of Texas/MD Anderson Cancer Center Dept of Onc., Houston, Texas
- Australia (3):
  - Pfizer Investigative Site 1003, North Sydney, New South Wales
  - Pfizer Investigative Site 1002, Westmead, New South Wales
  - Pfizer Investigator Site 1001, East Melbourne, Victoria
- Germany (4):
  - Pfizer Investigative Site 1050, Essen
  - Pfizer Investigative Site 1053, Gera
  - Pfizer Investigative Site 1052, Hanover
  - Pfizer Investigative Site 1051, München
- Pfizer Investigative Site 1101, Napoli, Italy
- Netherlands (2):
  - Pfizer Investigative Site 1151, Utrecht, The Netherlands
  - Pfizer Investigative Site 1150, Nijmegen

REFERENCES:
- [Derived] Schuler M, Zimmer L, Kim KB, Sosman JA, Ascierto PA, Postow MA, De Vos FYFL, van Herpen CML, Carlino MS, Johnson DB, Berking C, Reddy MB, Harney AS, Berlin JD, Amaria RN. Phase Ib/II Trial of Ribociclib in Combination with Binimetinib in Patients with NRAS-mutant Melanoma. Clin Cancer Res. 2022 Jul 15;28(14):3002-3010. doi: 10.1158/1078-0432.CCR-21-3872. PMID 35294522

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Upon study entry, all patients were required to provide either an archival tumor biopsy with the corresponding pathology report or a newly obtained tumor biopsy. Both parts of the study were limited to patients aged 18 or older with metastatic or locally advanced NRAS-mutant melanoma.
Pre-assignment Details: Screening details:
  Screening assessments were performed within 14 days prior to the first dose of ribociclib and binimetinib except for the pretreatment tumor biopsy, which was performed within 28 days before dosing. A total of 23 patients were screened but not enrolled.
Groups:
- Phase 1b 28-Day Schedule: A combined total of 61 patients were treated in the 28-day (n=29) and 21-day (n=32) treatment cycles, and all patients discontinued treatment. The starting dose in the 28-day schedule was binimetinib 45 mg BID + ribociclib 200 mg QD.
  28-Day Schedule: ribociclib was taken QD for 21 consecutive days followed by a 7-day planned break.
  Binimetinib was taken BID on a continuous dosing schedule.
- Phase 1b 21-Day Schedule: A combined total of 61 patients were treated in the 28-day (n=29) and 21-day (n=32) treatment cycles, and all patients discontinued treatment. The starting dose in the 21-day schedule was binimetinib 30 mg BID + ribociclib 200 mg QD.
  21-Day Schedule: ribociclib QD and binimetinib BID were taken QD for 14 consecutive days followed by a 7-day planned break.
- Phase 2 (Dose-expansion Phase): The dose-expansion phase was initiated with a newly recruited group of patients.
  A total of 41 patients were treated, and all patients (100%) discontinued treatment. Based on the recommendations of the dose-escalation meetings between the Sponsor and the Investigators, the RP2D and schedule for the combination of binimetinib and ribociclib to be used for the dose-expansion phase of the study was binimetinib 45 mg BID + ribociclib 200 mg QD on the 28-day schedule.
Period: MEK162 45mg BID+LEE011 200mg
Arm/Group | Phase 1b 28-Day Schedule | Phase 1b 21-Day Schedule | Phase 2 (Dose-expansion Phase)
Started | 16 | 6 | 41
Completed | 0 | 0 | 0
Not Completed | 16 | 6 | 41
Not completed — Adverse Event | 7 | 0 | 11
Not completed — Progressive disease | 8 | 6 | 23
Not completed — Withdrawal by Subject | 1 | 0 | 2
Not completed — Physician Decision | 0 | 0 | 4
Not completed — Death | 0 | 0 | 1
Period: MEK162 45mg BID+LEE011 250mg
Arm/Group | Phase 1b 28-Day Schedule | Phase 1b 21-Day Schedule | Phase 2 (Dose-expansion Phase)
Started | 3 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 3 | 0 | 0
Not completed — Progressive Disease | 2 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Period: MEK162 30mg BID+LEE011 300mg
Arm/Group | Phase 1b 28-Day Schedule | Phase 1b 21-Day Schedule | Phase 2 (Dose-expansion Phase)
Started | 4 | 2 | 0
Completed | 0 | 0 | 0
Not Completed | 4 | 2 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Progressive Disease | 3 | 2 | 0
Period: MEK162 45mg BID+LEE011 300mg
Arm/Group | Phase 1b 28-Day Schedule | Phase 1b 21-Day Schedule | Phase 2 (Dose-expansion Phase)
Started | 6 | 4 | 0
Completed | 0 | 0 | 0
Not Completed | 6 | 4 | 0
Not completed — Adverse Event | 1 | 1 | 0
Not completed — Progressive Disease | 4 | 3 | 0
Not completed — Death | 1 | 0 | 0
Period: MEK162 30mg LEE011 200mg
Arm/Group | Phase 1b 28-Day Schedule | Phase 1b 21-Day Schedule | Phase 2 (Dose-expansion Phase)
Started | 0 | 5 | 0
Completed | 0 | 0 | 0
Not Completed | 0 | 5 | 0
Not completed — Progressive Disease | 0 | 5 | 0
Period: MEK162 45mg LEE011 450mg
Arm/Group | Phase 1b 28-Day Schedule | Phase 1b 21-Day Schedule | Phase 2 (Dose-expansion Phase)
Started | 0 | 9 | 0
Completed | 0 | 0 | 0
Not Completed | 0 | 9 | 0
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Physician Decision | 0 | 2 | 0
Not completed — Progressive Disease | 0 | 6 | 0
Period: MEK162 45mg LEE011 600mg
Arm/Group | Phase 1b 28-Day Schedule | Phase 1b 21-Day Schedule | Phase 2 (Dose-expansion Phase)
Started | 0 | 6 | 0
Completed | 0 | 0 | 0
Not Completed | 0 | 6 | 0
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Progressive Disease | 0 | 5 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population consists of the Full Analysis Set (FAS), which includes all patients who received at least 1 dose of ribociclib or binimetinib.
Groups:
- Phase 1b 28-Day MEK162 45mg + LEE011 200mg: MEK162 45mg + LEE011 200mg
- Phase 1b 28-Day MEK162 45mg+LEE011 250mg: MEK162 45mg+LEE011 250mg
- Phase 1b 28-Day MEK162 30mg+LEE011 300mg; Phase 1b 21-Day MEK162 30mg+LEE011 300mg: MEK162 30mg+LEE011 300mg
- Phase 1b 28-Day MEK162 45mg+LEE011 300mg; Phase 1b 21-Day MEK162 45mg+LEE011 300mg: MEK162 45mg+LEE011 300mg
- Phase 1b 21-Day MEK162 30mg+LEE011 200mg: MEK162 30mg+LEE011 200mg
- Phase 1b 21-Day MEK162 45mg+LEE011 200mg; Phase 2: MEK162 45mg+LEE011 200mg: MEK162 45mg+LEE011 200mg
- Phase 1b 21-Day MEK162 45mg+LEE011 450mg: MEK162 45mg+LEE011 450mg
- Phase 1b 21-Day MEK162 45mg+LEE011 600mg: MEK162 45mg+LEE011 600mg
- Total: Total of all reporting groups
Arm/Group | Phase 1b 28-Day MEK162 45mg + LEE011 200mg | Phase 1b 28-Day MEK162 45mg+LEE011 250mg | Phase 1b 28-Day MEK162 30mg+LEE011 300mg | Phase 1b 28-Day MEK162 45mg+LEE011 300mg | Phase 1b 21-Day MEK162 30mg+LEE011 200mg | Phase 1b 21-Day MEK162 45mg+LEE011 200mg | Phase 1b 21-Day MEK162 30mg+LEE011 300mg | Phase 1b 21-Day MEK162 45mg+LEE011 300mg | Phase 1b 21-Day MEK162 45mg+LEE011 450mg | Phase 1b 21-Day MEK162 45mg+LEE011 600mg | Phase 2: MEK162 45mg+LEE011 200mg | Total
Number analyzed (Participants) | 16 | 3 | 4 | 6 | 5 | 6 | 2 | 4 | 9 | 6 | 41 | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 2 | 2 | 4 | 3 | 3 | 1 | 2 | 4 | 5 | 19 | 54
  >=65 years | 7 | 1 | 2 | 2 | 2 | 3 | 1 | 2 | 5 | 1 | 22 | 48
Age, Continuous [Median (Standard Deviation); unit: years] | 62 (14.51) | 57 (9.02) | 61.5 (21.30) | 56 (15.04) | 63.0 (7.50) | 62.5 (12.687) | 55.0 (18.38) | 63.5 (19.48) | 67.0 (8.59) | 58.5 (5.56) | 65 (12.35) | 61 (12.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 0 | 3 | 1 | 2 | 3 | 1 | 2 | 1 | 5 | 15 | 41
  Male | 8 | 3 | 1 | 5 | 3 | 3 | 1 | 2 | 8 | 1 | 26 | 61
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasian | 16 | 3 | 4 | 6 | 5 | 6 | 1 | 4 | 9 | 6 | 40 | 100
  Race: Other | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
Weight [Mean (Standard Deviation); unit: kilograms] | 82.57 (15.014) | 91.47 (20.093) | 71.30 (12.631) | 97.48 (35.464) | 73.66 (8.104) | 85.20 (20.733) | 80.80 (15.274) | 97.20 (24.554) | 92.41 (20.709) | 62.95 (6.111) | 79.63 (17.334) | 83.69 (20.621)
Body mass index [Mean (Standard Deviation); unit: (kg)/m^2] | 28.57 (5.136) | 26.84 (5.332) | 25.95 (3.347) | 30.38 (9.733) | 23.85 (2.451) | 27.80 (6.185) | 27.92 (7.526) | 31.71 (5.305) | 28.08 (6.594) | 23.50 (3.293) | 26.69 (5.014) | 27.34 (5.841)
ECOG performance status [Count of Participants; unit: Participants]
  0-Without restriction | 10 | 2 | 1 | 2 | 3 | 5 | 2 | 2 | 5 | 5 | 28 | 65
  1-Restricted in physically strenuous activity | 5 | 0 | 3 | 4 | 2 | 1 | 0 | 2 | 4 | 1 | 13 | 35
  2-Ambulatory and capable of all selfcare | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Dose Limiting Toxicities (Phase Ib)
Description: To estimate the maximum tolerate doses (MTDs) and/or identify the RP2D and schedule of LEE011 and MEK162 combination. A dose-limiting toxicity (DLT) was defined as an AE or clinically significant abnormal laboratory value assessed as unrelated to disease, disease progression, inter-current illness, or concomitant medications that occurred within the first cycle of treatment with ribociclib and binimetinib.
Time Frame: first 28 days of treatment
Population: Analysis is comprised of the dose-determining set, which is all patients from the safety set who either met the minimum exposure criterion below and had sufficient safety evaluations during Cycle 1 or discontinued earlier due to DLT during Cycle 1.
Measure: Number; unit: occurrence
Arm/Group | Phase 1b 28-Day MEK162 45mg + LEE011 200mg | Phase 1b 28-Day MEK162 45mg+LEE011 250mg | Phase 1b 28-Day MEK162 30mg+LEE011 300mg | Phase 1b 28-Day MEK162 45mg+LEE011 300mg | Phase 1b 21-Day MEK162 30mg+LEE011 200mg | Phase 1b 21-Day MEK162 45mg+LEE011 200mg | Phase 1b 21-Day MEK162 30mg+LEE011 300mg | Phase 1b 21-Day MEK162 45mg+LEE011 300mg | Phase 1b 21-Day MEK162 45mg+LEE011 450mg | Phase 1b 21-Day MEK162 45mg+LEE011 600mg
Number analyzed (Participants) | 16 | 3 | 4 | 6 | 5 | 6 | 2 | 4 | 9 | 6
occurrence | 2 | 0 | 1 | 3 | 0 | 1 | 0 | 1 | 2 | 0

2. Primary Outcome: Objective Response Rate (ORR) (Phase II)
Description: ORR is the proportion of patients with best overall response of complete response (CR) or partial response (PR) by month 2 assessed according to RECIST 1.1 criteria. ORR is done to describe the anti-tumor activity of LEE011 and MEK162 combination. The primary analysis of the ORR was based on the Investigator's assessment of overall lesion responses per RECIST 1.1.
Time Frame: Approximately 12 months after the FPFV
Population: Analysis population consist of the Full Analysis Set, which included all patients who received at least one dose of binimetinib or ribociclib and was used for the analysis of all endpoints unless noted otherwise.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 2: Dose Expansion: binimetinib 45 mg BID + ribociclib 200 mg QD (MEK 45mg + LEE 200mg)
Arm/Group | Phase 2: Dose Expansion
Number analyzed (Participants) | 41
Participants | 8

3. Secondary Outcome: Plasma Concentration-time Profile (AUCtau) of LEE011 (Phase Ib)
Description: To Characterize the PK profiles of LEE011 as well as any other significant metabolites identified (Phase Ib).
Time Frame: Cycle 1 Day 1
Population: Analysis population consist of the pharmacokinetic analysis set (PAS) which consisted of all patients who had at least one blood sample providing evaluable PK data and received at least one dose of study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/ml
Arm/Group | Phase 1b 28-Day MEK162 45mg + LEE011 200mg | Phase 1b 28-Day MEK162 45mg+LEE011 250mg | Phase 1b 28-Day MEK162 30mg+LEE011 300mg | Phase 1b 28-Day MEK162 45mg+LEE011 300mg | Phase 1b 21-Day MEK162 30mg+LEE011 200mg | Phase 1b 21-Day MEK162 45mg+LEE011 200mg | Phase 1b 21-Day MEK162 30mg+LEE011 300mg | Phase 1b 21-Day MEK162 45mg+LEE011 300mg | Phase 1b 21-Day MEK162 45mg+LEE011 450mg | Phase 1b 21-Day MEK162 45mg+LEE011 600mg
Number analyzed (Participants) | 15 | 3 | 4 | 6 | 4 | 5 | 1 | 4 | 9 | 5
h*ng/ml | 2120 (66.2) | 3020 (99.4) | 5280 (27.8) | 3860 (42.3) | 2340 (113) | 2230 (74.5) | 5020 (NA) — Insufficient number of participants to calculate. | 2960 (46.4) | 5550 (50.3) | 9840 (65.7)

4. Secondary Outcome: Plasma Concentration-time Profile (AUCtau) of MEK162 (Phase Ib)
Description: To Characterize the PK profiles of MEK162 as well as any other significant metabolites identified (Phase Ib).
Time Frame: Cycle 1 Day 1
Population: The analysis group is comprised of the pharmacokinetic analysis set (PAS) consisted of all patients who had at least one blood sample providing evaluable PK data and received at least one dose of study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/ml
Arm/Group | Phase 1b 28-Day MEK162 45mg + LEE011 200mg | Phase 1b 28-Day MEK162 45mg+LEE011 250mg | Phase 1b 28-Day MEK162 30mg+LEE011 300mg | Phase 1b 28-Day MEK162 45mg+LEE011 300mg | Phase 1b 21-Day MEK162 30mg+LEE011 200mg | Phase 1b 21-Day MEK162 45mg+LEE011 200mg | Phase 1b 21-Day MEK162 30mg+LEE011 300mg | Phase 1b 21-Day MEK162 45mg+LEE011 300mg | Phase 1b 21-Day MEK162 45mg+LEE011 450mg | Phase 1b 21-Day MEK162 45mg+LEE011 600mg
Number analyzed (Participants) | 6 | 1 | 1 | 1 | 2 | 3 | 2 | 1 | 2 | 1
h*ng/ml | 1310 (36.8) | 1070 (NA) — Insufficient number of participants to calculate. | 1640 (NA) — Insufficient number of participants to calculate. | 1240 (NA) — Insufficient number of participants to calculate. | 1610 (76) | 1820 (82.1) | 747 (31.8) | 2740 (NA) — Insufficient number of participants to calculate. | 2110 (44.2) | 4060 (NA) — Insufficient number of participants to calculate.

5. Secondary Outcome: Plasma Concentration-time Profile (AUCtau,ss) of LEE011 (Phase Ib)
Description: To Characterize the PK profiles of LEE011 as well as any other significant metabolites identified (Phase Ib).
Time Frame: For the 28-day schedule the steady-state parameter time frame was Cycle 1 Day 21, and for the 21-day schedule the steady-state parameter time frame was Cycle 1 Day 14
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Phase 1b 28-Day MEK162 45mg + LEE011 200mg | Phase 1b 28-Day MEK162 45mg+LEE011 250mg | Phase 1b 28-Day MEK162 30mg+LEE011 300mg | Phase 1b 28-Day MEK162 45mg+LEE011 300mg | Phase 1b 21-Day MEK162 30mg+LEE011 200mg | Phase 1b 21-Day MEK162 45mg+LEE011 200mg | Phase 1b 21-Day MEK162 30mg+LEE011 300mg | Phase 1b 21-Day MEK162 45mg+LEE011 300mg | Phase 1b 21-Day MEK162 45mg+LEE011 450mg | Phase 1b 21-Day MEK162 45mg+LEE011 600mg
Number analyzed (Participants) | 13 | 1 | 1 | 2 | 4 | 5 | 2 | 2 | 5 | 5
h*ng/mL | 3080 (63.2) | 15000 (NA) — Insufficient number of participants to calculate. | 8650 (NA) — Insufficient number of participants to calculate. | 7050 (41.3) | 4700 (28.9) | 4370 (60.3) | 7480 (2.89) | 9570 (50.5) | 11100 (29.1) | 30700 (46.4)

6. Secondary Outcome: Plasma Concentration-time Profile (AUCtau,ss) of MEK162 (Phase Ib)
Description: To Characterize the PK profiles of MEK162 as well as any other significant metabolites identified (Phase Ib).
Time Frame: as for outcome 5
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Phase 1b 28-Day MEK162 45mg + LEE011 200mg | Phase 1b 28-Day MEK162 45mg+LEE011 250mg | Phase 1b 28-Day MEK162 30mg+LEE011 300mg | Phase 1b 28-Day MEK162 45mg+LEE011 300mg | Phase 1b 21-Day MEK162 30mg+LEE011 200mg | Phase 1b 21-Day MEK162 45mg+LEE011 200mg | Phase 1b 21-Day MEK162 30mg+LEE011 300mg | Phase 1b 21-Day MEK162 45mg+LEE011 300mg | Phase 1b 21-Day MEK162 45mg+LEE011 450mg | Phase 1b 21-Day MEK162 45mg+LEE011 600mg
Number analyzed (Participants) | 11 | 1 | 0 | 4 | 4 | 4 | 2 | 3 | 4 | 5
h*ng/mL | 2250 (37.7) | 2450 (NA) — Insufficient number of participants to calculate. |  | 1540 (30.0) | 2180 (12.1) | 2980 (58.9) | 1990 (22.2) | 3680 (40.9) | 2840 (57.5) | 3340 (86.5)

7. Secondary Outcome: Plasma Concentration-time Profile (Cmin,ss) of LEE011 (Phase Ib)
Description: To Characterize the PK profiles of LEE011 as well as any other significant metabolites identified (Phase Ib).
Time Frame: For the 28-day schedule the steady-state parameter time frame was predose on Cycle 1 Day 21, and for the 21-day schedule the steady-state parameter time frame was predose on Cycle 1 Day 14
Population: Analysis population consist of the pharmacokinetic analysis set (PAS), which consisted of all patients who had at least one blood sample providing evaluable PK data and received at least one dose of study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase 1b 28-Day MEK162 45mg + LEE011 200mg | Phase 1b 28-Day MEK162 45mg+LEE011 250mg | Phase 1b 28-Day MEK162 30mg+LEE011 300mg | Phase 1b 28-Day MEK162 45mg+LEE011 300mg | Phase 1b 21-Day MEK162 30mg+LEE011 200mg | Phase 1b 21-Day MEK162 45mg+LEE011 200mg | Phase 1b 21-Day MEK162 30mg+LEE011 300mg | Phase 1b 21-Day MEK162 45mg+LEE011 300mg | Phase 1b 21-Day MEK162 45mg+LEE011 450mg | Phase 1b 21-Day MEK162 45mg+LEE011 600mg
Number analyzed (Participants) | 14 | 2 | 1 | 4 | 4 | 5 | 2 | 2 | 5 | 6
ng/mL | 88.1 (56.3) | 256 (79.8) | 220 (NA) — Insufficient number of participants to calculate. | 113 (56.4) | 117 (39.8) | 97.6 (77.8) | 140 (25.6) | 216 (7.88) | 264 (44.9) | 570 (91.3)

8. Secondary Outcome: Plasma Concentration-time Profile (Cmin,ss) of MEK162 (Phase Ib)
Description: To Characterize the PK profiles of MEK162 as well as any other significant metabolites identified (Phase Ib).
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase 1b 28-Day MEK162 45mg + LEE011 200mg | Phase 1b 28-Day MEK162 45mg+LEE011 250mg | Phase 1b 28-Day MEK162 30mg+LEE011 300mg | Phase 1b 28-Day MEK162 45mg+LEE011 300mg | Phase 1b 21-Day MEK162 30mg+LEE011 200mg | Phase 1b 21-Day MEK162 45mg+LEE011 200mg | Phase 1b 21-Day MEK162 30mg+LEE011 300mg | Phase 1b 21-Day MEK162 45mg+LEE011 300mg | Phase 1b 21-Day MEK162 45mg+LEE011 450mg | Phase 1b 21-Day MEK162 45mg+LEE011 600mg
Number analyzed (Participants) | 11 | 2 | 1 | 3 | 4 | 4 | 1 | 3 | 4 | 6
ng/mL | 73.2 (75.4) | 188 (73.9) | 84.2 (NA) — Insufficient number of participants to calculate. | 43.9 (60.7) | 103 (31.4) | 90.4 (20.0) | 123 (NA) — Insufficient number of participants to calculate. | 178 (38.1) | 63.9 (94.3) | 179 (98.3)

9. Secondary Outcome: Plasma Concentration-time Profile (Cmax) of LEE011 (Phase Ib)
Description: To Characterize the PK profiles of LEE011 as well as any other significant metabolites identified (Phase Ib).
Time Frame: Cycle 1 Day 1
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase 1b 28-Day MEK162 45mg + LEE011 200mg | Phase 1b 28-Day MEK162 45mg+LEE011 250mg | Phase 1b 28-Day MEK162 30mg+LEE011 300mg | Phase 1b 28-Day MEK162 45mg+LEE011 300mg | Phase 1b 21-Day MEK162 30mg+LEE011 200mg | Phase 1b 21-Day MEK162 45mg+LEE011 200mg | Phase 1b 21-Day MEK162 30mg+LEE011 300mg | Phase 1b 21-Day MEK162 45mg+LEE011 300mg | Phase 1b 21-Day MEK162 45mg+LEE011 450mg | Phase 1b 21-Day MEK162 45mg+LEE011 600mg
Number analyzed (Participants) | 15 | 3 | 4 | 6 | 4 | 5 | 1 | 4 | 9 | 5
ng/mL | 217 (90.5) | 271 (87.4) | 555 (44.4) | 374 (47.9) | 236 (143) | 229 (86.0) | 368 (NA) — Insufficient number of participants to calculate. | 307 (33.0) | 506 (65.6) | 1030 (54.1)

10. Secondary Outcome: Plasma Concentration-time Profile (Cmax) of MEK162 (Phase Ib)
Description: To Characterize the PK profiles of MEK162 as well as any other significant metabolites identified (Phase Ib).
Time Frame: Cycle 1 Day 1
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase 1b 28-Day MEK162 45mg + LEE011 200mg | Phase 1b 28-Day MEK162 45mg+LEE011 250mg | Phase 1b 28-Day MEK162 30mg+LEE011 300mg | Phase 1b 28-Day MEK162 45mg+LEE011 300mg | Phase 1b 21-Day MEK162 30mg+LEE011 200mg | Phase 1b 21-Day MEK162 45mg+LEE011 200mg | Phase 1b 21-Day MEK162 30mg+LEE011 300mg | Phase 1b 21-Day MEK162 45mg+LEE011 300mg | Phase 1b 21-Day MEK162 45mg+LEE011 450mg | Phase 1b 21-Day MEK162 45mg+LEE011 600mg
Number analyzed (Participants) | 15 | 3 | 3 | 6 | 5 | 6 | 2 | 4 | 9 | 5
ng/mL | 315 (55.7) | 296 (48.4) | 247 (59.7) | 231 (47.3) | 234 (73.9) | 453 (67.1) | 163 (47.8) | 396 (52.7) | 385 (50.3) | 402 (69.8)

11. Secondary Outcome: Plasma Concentration-time Profile (Cmax,ss) of LEE011 (Phase Ib)
Description: To Characterize the PK profiles of LEE011 as well as any other significant metabolites identified (Phase Ib).
Time Frame: as for outcome 5
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase 1b 28-Day MEK162 45mg + LEE011 200mg | Phase 1b 28-Day MEK162 45mg+LEE011 250mg | Phase 1b 28-Day MEK162 30mg+LEE011 300mg | Phase 1b 28-Day MEK162 45mg+LEE011 300mg | Phase 1b 21-Day MEK162 30mg+LEE011 200mg | Phase 1b 21-Day MEK162 45mg+LEE011 200mg | Phase 1b 21-Day MEK162 30mg+LEE011 300mg | Phase 1b 21-Day MEK162 45mg+LEE011 300mg | Phase 1b 21-Day MEK162 45mg+LEE011 450mg | Phase 1b 21-Day MEK162 45mg+LEE011 600mg
Number analyzed (Participants) | 14 | 2 | 1 | 4 | 5 | 5 | 2 | 2 | 5 | 6
ng/mL | 220 (76.5) | 343 (150) | 220 (NA) — Insufficient number of participants to calculate. | 530 (30.6) | 373 (62.4) | 341 (69.0) | 543 (11.9) | 747 (33.0) | 727 (34.7) | 1910 (38.5)

12. Secondary Outcome: Plasma Concentration-time Profile (Cmax,ss) of MEK162 (Phase Ib)
Description: To Characterize the PK profiles of MEK162 as well as any other significant metabolites identified (Phase Ib).
Time Frame: as for outcome 5
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase 1b 28-Day MEK162 45mg + LEE011 200mg | Phase 1b 28-Day MEK162 45mg+LEE011 250mg | Phase 1b 28-Day MEK162 30mg+LEE011 300mg | Phase 1b 28-Day MEK162 45mg+LEE011 300mg | Phase 1b 21-Day MEK162 30mg+LEE011 200mg | Phase 1b 21-Day MEK162 45mg+LEE011 200mg | Phase 1b 21-Day MEK162 30mg+LEE011 300mg | Phase 1b 21-Day MEK162 45mg+LEE011 300mg | Phase 1b 21-Day MEK162 45mg+LEE011 450mg | Phase 1b 21-Day MEK162 45mg+LEE011 600mg
Number analyzed (Participants) | 11 | 2 | 0 | 4 | 5 | 4 | 2 | 3 | 4 | 6
ng/mL | 441 (52.6) | 309 (1.60) |  | 284 (14.5) | 376 (18.0) | 444 (36.6) | 367 (31.5) | 590 (12.3) | 452 (59.2) | 471 (75.6)

13. Secondary Outcome: Plasma Concentration-time Profile (Tmax) of LEE011 (Phase Ib)
Description: To Characterize the PK profiles of LEE011 as well as any other significant metabolites identified (Phase Ib).
Time Frame: Cycle 1 Day 1
Population: as for outcome 7
Measure: Median (Full Range); unit: h
Arm/Group | Phase 1b 28-Day MEK162 45mg + LEE011 200mg | Phase 1b 28-Day MEK162 45mg+LEE011 250mg | Phase 1b 28-Day MEK162 30mg+LEE011 300mg | Phase 1b 28-Day MEK162 45mg+LEE011 300mg | Phase 1b 21-Day MEK162 30mg+LEE011 200mg | Phase 1b 21-Day MEK162 45mg+LEE011 200mg | Phase 1b 21-Day MEK162 30mg+LEE011 300mg | Phase 1b 21-Day MEK162 45mg+LEE011 300mg | Phase 1b 21-Day MEK162 45mg+LEE011 450mg | Phase 1b 21-Day MEK162 45mg+LEE011 600mg
Number analyzed (Participants) | 15 | 3 | 4 | 6 | 4 | 5 | 1 | 4 | 9 | 5
h | 2.12 [1.00 to 24.92] | 3.75 [2.12 to 4.10] | 2.98 [0.67 to 4.08] | 1.50 [0.52 to 4.00] | 2.98 [1.98 to 7.95] | 1.12 [0.87 to 3.83] | 4.22 [4.22 to 4.22] | 1.50 [1.00 to 8.00] | 2.13 [1.00 to 4.03] | 2.03 [1.62 to 2.13]

14. Secondary Outcome: Plasma Concentration-time Profile (Tmax) of MEK162 (Phase Ib)
Description: To Characterize the PK profiles of MEK162 as well as any other significant metabolites identified (Phase Ib).
Time Frame: Cycle 1 Day 1
Population: as for outcome 7
Measure: Median (Full Range); unit: h
Arm/Group | Phase 1b 28-Day MEK162 45mg + LEE011 200mg | Phase 1b 28-Day MEK162 45mg+LEE011 250mg | Phase 1b 28-Day MEK162 30mg+LEE011 300mg | Phase 1b 28-Day MEK162 45mg+LEE011 300mg | Phase 1b 21-Day MEK162 30mg+LEE011 200mg | Phase 1b 21-Day MEK162 45mg+LEE011 200mg | Phase 1b 21-Day MEK162 30mg+LEE011 300mg | Phase 1b 21-Day MEK162 45mg+LEE011 300mg | Phase 1b 21-Day MEK162 45mg+LEE011 450mg | Phase 1b 21-Day MEK162 45mg+LEE011 600mg
Number analyzed (Participants) | 15 | 3 | 3 | 6 | 5 | 6 | 2 | 4 | 9 | 5
h | 1.08 [0.85 to 8.00] | 2.05 [0.50 to 2.12] | 1.02 [1.00 to 1.97] | 2.00 [.52 to 4.00] | 1.98 [0.43 to 7.95] | 1.11 [0.87 to 2.05] | 0.76 [0.52 to 1.00] | 2.00 [1.00 to 4.15] | 2.17 [1.00 to 8.08] | 1.17 [0.47 to 4.02]

15. Secondary Outcome: Plasma Concentration-time Profile (Tmax,ss) of LEE011 (Phase Ib)
Description: To Characterize the PK profiles of LEE011 as well as any other significant metabolites identified (Phase Ib).
Time Frame: as for outcome 5
Population: as for outcome 7
Measure: Median (Full Range); unit: h
Arm/Group | Phase 1b 28-Day MEK162 45mg + LEE011 200mg | Phase 1b 28-Day MEK162 45mg+LEE011 250mg | Phase 1b 28-Day MEK162 30mg+LEE011 300mg | Phase 1b 28-Day MEK162 45mg+LEE011 300mg | Phase 1b 21-Day MEK162 30mg+LEE011 200mg | Phase 1b 21-Day MEK162 45mg+LEE011 200mg | Phase 1b 21-Day MEK162 30mg+LEE011 300mg | Phase 1b 21-Day MEK162 45mg+LEE011 300mg | Phase 1b 21-Day MEK162 45mg+LEE011 450mg | Phase 1b 21-Day MEK162 45mg+LEE011 600mg
Number analyzed (Participants) | 14 | 2 | 1 | 4 | 5 | 5 | 2 | 2 | 5 | 6
h | 2.25 [0.00 to 7.5] | 5.90 [4.00 to 7.80] | 23.93 [23.93 to 23.93] | 2.99 [2.00 to 4.00] | 4.00 [1.03 to 7.87] | 1.87 [0.50 to 4.08] | 2.03 [1.93 to 2.12] | 4.05 [2.08 to 6.02] | 3.92 [2.08 to 4.13] | 1.93 [1.02 to 4.00]

16. Secondary Outcome: Plasma Concentration-time Profile (Tmax,ss) of MEK162 (Phase Ib)
Description: To Characterize the PK profiles of MEK162 as well as any other significant metabolites identified (Phase Ib).
Time Frame: as for outcome 5
Population: as for outcome 7
Measure: Median (Full Range); unit: h
Arm/Group | Phase 1b 28-Day MEK162 45mg + LEE011 200mg | Phase 1b 28-Day MEK162 45mg+LEE011 250mg | Phase 1b 28-Day MEK162 30mg+LEE011 300mg | Phase 1b 28-Day MEK162 45mg+LEE011 300mg | Phase 1b 21-Day MEK162 30mg+LEE011 200mg | Phase 1b 21-Day MEK162 45mg+LEE011 200mg | Phase 1b 21-Day MEK162 30mg+LEE011 300mg | Phase 1b 21-Day MEK162 45mg+LEE011 300mg | Phase 1b 21-Day MEK162 45mg+LEE011 450mg | Phase 1b 21-Day MEK162 45mg+LEE011 600mg
Number analyzed (Participants) | 11 | 2 | 0 | 4 | 5 | 4 | 2 | 3 | 4 | 6
h | 1.00 [0.75 to 4.03] | 3.03 [1.97 to 4.10] |  | 2.31 [1.00 to 4.00] | 1.00 [0.53 to 4.13] | 1.96 [1.00 to 3.95] | 1.49 [1.05 to 1.93] | 2.02 [1.08 to 6.02] | 1.92 [0.98 to 2.08] | 1.49 [0.00 to 3.63]

17. Secondary Outcome: Plasma Concentration-time Profile (Accumulation Ratio, Racc_AUC) of LEE011 (Phase Ib)
Description: To Characterize the PK profiles of LEE011 as well as any other significant metabolites identified (Phase Ib).
Time Frame: as for outcome 5
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (hr*ng/mL) / (hr*ng/mL)
Arm/Group | Phase 1b 28-Day MEK162 45mg + LEE011 200mg | Phase 1b 28-Day MEK162 45mg+LEE011 250mg | Phase 1b 28-Day MEK162 30mg+LEE011 300mg | Phase 1b 28-Day MEK162 45mg+LEE011 300mg | Phase 1b 21-Day MEK162 30mg+LEE011 200mg | Phase 1b 21-Day MEK162 45mg+LEE011 200mg | Phase 1b 21-Day MEK162 30mg+LEE011 300mg | Phase 1b 21-Day MEK162 45mg+LEE011 300mg | Phase 1b 21-Day MEK162 45mg+LEE011 450mg | Phase 1b 21-Day MEK162 45mg+LEE011 600mg
Number analyzed (Participants) | 13 | 1 | 1 | 4 | 4 | 5 | 2 | 2 | 5 | 5
(hr*ng/mL) / (hr*ng/mL) | 1.51 (53.9) | 2.52 (NA) — Insufficient number of participants to calculate. | 2.25 (NA) — Insufficient number of participants to calculate. | 2.29 (38.4) | 2.89 (32.8) | 2.28 (54.6) | 3.29 (165) | 3.50 (8.68) | 1.97 (45.4) | 3.95 (58.6)

18. Secondary Outcome: Plasma Concentration-time Profile (Accumulation Ratio, Racc_AUC) of MEK162 (Phase Ib)
Description: To Characterize the PK profiles of MEK162 as well as any other significant metabolites identified (Phase Ib).
Time Frame: as for outcome 5
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (hr*ng/mL) / (hr*ng/mL
Arm/Group | Phase 1b 28-Day MEK162 45mg + LEE011 200mg | Phase 1b 28-Day MEK162 45mg+LEE011 250mg | Phase 1b 28-Day MEK162 30mg+LEE011 300mg | Phase 1b 28-Day MEK162 45mg+LEE011 300mg | Phase 1b 21-Day MEK162 30mg+LEE011 200mg | Phase 1b 21-Day MEK162 45mg+LEE011 200mg | Phase 1b 21-Day MEK162 30mg+LEE011 300mg | Phase 1b 21-Day MEK162 45mg+LEE011 300mg | Phase 1b 21-Day MEK162 45mg+LEE011 450mg | Phase 1b 21-Day MEK162 45mg+LEE011 600mg
Number analyzed (Participants) | 13 | 1 | 1 | 4 | 4 | 5 | 2 | 2 | 5 | 5
(hr*ng/mL) / (hr*ng/mL | 2.53 (45.8) | 7.59 (NA) — Insufficient number of participants to calculate. | 1.74 (NA) — Insufficient number of participants to calculate. | 3.39 (15.2) | 4.47 (21.5) | 2.26 (27.3) | 3.14 (161) | 3.48 (53.0) | 2.09 (53.5) | 3.06 (26.0)

19. Secondary Outcome: Plasma Concentration-time Profile (T1/2,ss) of LEE011 (Phase Ib)
Description: To Characterize the PK profiles of LEE011 as well as any other significant metabolites identified (Phase Ib).
Time Frame: as for outcome 5
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Phase 1b 28-Day MEK162 45mg + LEE011 200mg | Phase 1b 28-Day MEK162 45mg+LEE011 250mg | Phase 1b 28-Day MEK162 30mg+LEE011 300mg | Phase 1b 28-Day MEK162 45mg+LEE011 300mg | Phase 1b 21-Day MEK162 30mg+LEE011 200mg | Phase 1b 21-Day MEK162 45mg+LEE011 200mg | Phase 1b 21-Day MEK162 30mg+LEE011 300mg | Phase 1b 21-Day MEK162 45mg+LEE011 300mg | Phase 1b 21-Day MEK162 45mg+LEE011 450mg | Phase 1b 21-Day MEK162 45mg+LEE011 600mg
Number analyzed (Participants) | 11 | 1 | 1 | 4 | 4 | 5 | 2 | 2 | 4 | 5
h | 16.7 (83.6) | 32.9 (NA) — Insufficient number of participants to calculate. | 28.2 (NA) — Insufficient number of participants to calculate. | 28.0 (54.7) | 38.5 (44.4) | 26.9 (82.0) | 275 (64.5) | 49.5 (10.3) | 30.3 (17.6) | 55.3 (73.1)

20. Secondary Outcome: Plasma Concentration-time Profile (T1/2,ss) of MEK162 (Phase Ib)
Description: To Characterize the PK profiles of MEK162 as well as any other significant metabolites identified (Phase Ib).
Time Frame: as for outcome 5
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Phase 1b 28-Day MEK162 45mg + LEE011 200mg | Phase 1b 28-Day MEK162 45mg+LEE011 250mg | Phase 1b 28-Day MEK162 30mg+LEE011 300mg | Phase 1b 28-Day MEK162 45mg+LEE011 300mg | Phase 1b 21-Day MEK162 30mg+LEE011 200mg | Phase 1b 21-Day MEK162 45mg+LEE011 200mg | Phase 1b 21-Day MEK162 30mg+LEE011 300mg | Phase 1b 21-Day MEK162 45mg+LEE011 300mg | Phase 1b 21-Day MEK162 45mg+LEE011 450mg | Phase 1b 21-Day MEK162 45mg+LEE011 600mg
Number analyzed (Participants) | 11 | 2 | 0 | 4 | 4 | 4 | 2 | 3 | 4 | 5
h | 8.17 (30.6) | 7.38 (92.6) |  | 6.33 (81.1) | 15.0 (54.8) | 5.21 (73.2) | 15.4 (11.4) | 8.95 (23.9) | 8.73 (19.3) | 12.0 (31.2)

21. Secondary Outcome: Plasma Concentration-time Profile (CL/F) of LEE011 (Phase Ib)
Description: To Characterize the PK profiles of LEE011 as well as any other significant metabolites identified (Phase Ib).
Time Frame: Cycle 1 Day 1
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Phase 1b 28-Day MEK162 45mg + LEE011 200mg | Phase 1b 28-Day MEK162 45mg+LEE011 250mg | Phase 1b 28-Day MEK162 30mg+LEE011 300mg | Phase 1b 28-Day MEK162 45mg+LEE011 300mg | Phase 1b 21-Day MEK162 30mg+LEE011 200mg | Phase 1b 21-Day MEK162 45mg+LEE011 200mg | Phase 1b 21-Day MEK162 30mg+LEE011 300mg | Phase 1b 21-Day MEK162 45mg+LEE011 300mg | Phase 1b 21-Day MEK162 45mg+LEE011 450mg | Phase 1b 21-Day MEK162 45mg+LEE011 600mg
Number analyzed (Participants) | 8 | 1 | 2 | 5 | 2 | 3 | 0 | 3 | 4 | 5
L/h | 72.7 (75.4) | 41.2 (NA) — Insufficient number of participants to calculate. | 39.2 (26.7) | 67.6 (35.9) | 34.3 (81.7) | 57.2 (52.7) |  | 93.9 (36.1) | 78.4 (16.0) | 48.7 (68.8)

22. Secondary Outcome: Plasma Concentration-time Profile (CL/F) of MEK162 (Phase Ib)
Description: To Characterize the PK profiles of MEK162 as well as any other significant metabolites identified (Phase Ib).
Time Frame: Cycle 1 Day 1
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Phase 1b 28-Day MEK162 45mg + LEE011 200mg | Phase 1b 28-Day MEK162 45mg+LEE011 250mg | Phase 1b 28-Day MEK162 30mg+LEE011 300mg | Phase 1b 28-Day MEK162 45mg+LEE011 300mg | Phase 1b 21-Day MEK162 30mg+LEE011 200mg | Phase 1b 21-Day MEK162 45mg+LEE011 200mg | Phase 1b 21-Day MEK162 30mg+LEE011 300mg | Phase 1b 21-Day MEK162 45mg+LEE011 300mg | Phase 1b 21-Day MEK162 45mg+LEE011 450mg | Phase 1b 21-Day MEK162 45mg+LEE011 600mg
Number analyzed (Participants) | 6 | 1 | 1 | 1 | 2 | 3 | 2 | 1 | 2 | 1
L/h | 32.5 (36.3) | 35.9 (NA) — Insufficient number of participants to calculate. | 17.8 (NA) — Insufficient number of participants to calculate. | 35.5 (NA) — Insufficient number of participants to calculate. | 17.9 (80.7) | 23.9 (83.6) | 37.2 (23.0) | 15.9 (NA) — Insufficient number of participants to calculate. | 20.8 (45.8) | 10.2 (NA) — Insufficient number of participants to calculate.

23. Secondary Outcome: Number of Participants With Adverse Drug Reactions
Description: Safety and tolerability will be characterized through the incidence and severity of adverse drug reactions, serious adverse drug reactions, changes in hematology and chemistry values, vital signs, electrocardiograms (ECGs), dose interruptions, dose reduction and dose intensity.
Time Frame: Approximately 12 months after FPFV
Population: Analysis group consists of the safety set, which included all patients who received at least 1 dose of ribociclib or binimetinib and had at least 1 postbaseline safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b 28-Day MEK162 45mg + LEE011 200mg | Phase 1b 28-Day MEK162 45mg+LEE011 250mg | Phase 1b 28-Day MEK162 30mg+LEE011 300mg | Phase 1b 28-Day MEK162 45mg+LEE011 300mg | Phase 1b 21-Day MEK162 30mg+LEE011 200mg | Phase 1b 21-Day MEK162 45mg+LEE011 200mg | Phase 1b 21-Day MEK162 30mg+LEE011 300mg | Phase 1b 21-Day MEK162 45mg+LEE011 300mg | Phase 1b 21-Day MEK162 45mg+LEE011 450mg | Phase 1b 21-Day MEK162 45mg+LEE011 600mg | Phase 2: MEK162 45mg+LEE011 200mg
Number analyzed (Participants) | 16 | 3 | 4 | 6 | 5 | 6 | 2 | 4 | 9 | 6 | 41
Participants | 16 | 3 | 4 | 6 | 5 | 6 | 2 | 4 | 9 | 6 | 41

24. Secondary Outcome: Duration of Response (DoR) - Phase 2
Description: To assess clinical safety as per RECIST 1.1. Evaluation will occur continuously throughout the trial until progression, or death due to underlying cancer.
  Please note: As clinicaltrials.gov only allows numerical data entry, the value of 999 indicates "not estimable" for confidence interval.
Time Frame: Approximately 12 months after the FPFV
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Phase 2: Dose Expansion: The dose-expansion phase was initiated with a newly recruited group of patients.
  Binimetinib 45 mg BID + ribociclib 200 mg QD on 28-day schedule
Arm/Group | Phase 2: Dose Expansion
Number analyzed (Participants) | 41
months | 10.3 [4.1 to 999]

25. Secondary Outcome: Time to Progression (TTP) - Phase 2
Description: To assess clinical safety as per RECIST 1.1. Evaluation will occur continuously throughout the trial until progression, or death due to underlying cancer.
Time Frame: Approximately 12 months after the FPFV
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: Dose Expansion
Number analyzed (Participants) | 41
months | 3.7 [3.5 to 5.6]

26. Secondary Outcome: Progression Free Survival (PFS) - Phase 1b and Phase 2
Description: To assess clinical safety as per RECIST 1.1. Evaluation will occur continuously throughout the trial until progression, or death due to underlying cancer.
  In the Phase 1b part, patients were combined for purposes of PFS analyses based on schedule received, since too few patients received any individual dose level to allow for valid PFS estimates within the respective dose levels. This is how the data were analyses and presented for the clinical study report.
Time Frame: Approximately 12 months after the FPFV
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1b 28-Day Schedule | Phase 1b 21-Day Schedule | Phase 2 (Dose-expansion Phase)
Number analyzed (Participants) | 29 | 32 | 41
months | 6.7 [3.5 to 9.2] | 4.1 [2.8 to 6.1] | 3.7 [3.5 to 5.6]

27. Secondary Outcome: Overall Survival (OS) - Phase ll
Description: as for outcome 25
Time Frame: Approximately 12 months after the FPFV
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: Dose Expansion
Number analyzed (Participants) | 41
months | 11.3 [9.3 to 14.2]

28. Secondary Outcome: Best Overall Response (BOR) - Phase II
Description: To assess clinical safety according to RECIST 1.1. Evaluation will occur continuously throughout the trial until progression, or death due to underlying cancer.
Time Frame: Approximately 12 months after the FPFV
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Dose Expansion
Number analyzed (Participants) | 41
Participants
  Complete Response | 0
  Partial Response | 8
  Stable Disease | 21
  Progressive Disease | 6
  Non-CR/Non-PD | 0
  Unknown | 6

ADVERSE EVENTS:
Time Frame: Adverse Events (AE) were collected during the study, which began in June 2013 and concluded February 2018. After signing of the informed consent until 30 days after study treatment discontinuation.
Description: An AE is defined as the appearance of (or worsening of any pre-existing) undesirable sign(s), symptom(s), or medical condition(s) that occur after patient's signed informed consent has been obtained.
Groups:
- Phase 1b - 28 Day MEK162 45mg+LEE011 200mg; Phase 1b - 21 Day MEK162 45mg+LEE011 200mg: MEK162 45mg BID+LEE011 200mg QD
- Phase 1b - 28 Day MEK162 45mg+LEE011 250mg: MEK162 45mg BID+LEE011 250mg QD
- Phase 1b - 28 Day MEK162 30mg+LEE011 300mg; Phase 1b - 21 Day MEK162 30mg+LEE011 300mg: MEK162 30mg BID+LEE011 300mg QD
- Phase 1b - 28 Day MEK162 45mg+LEE011 300mg; Phase 1b - 21 Day MEK162 45mg+LEE011 300mg: MEK162 45mg BID+LEE011 300mg QD
- Phase 1b - 21 Day MEK162 30mg+LEE011 200mg: MEK162 30mg BID+LEE011 200mg QD
- Phase 1b - 21 Day MEK162 45mg+LEE011 450mg: MEK162 45mg BID+LEE011 450mg QD
- Phase 1b - 21 Day MEK162 45mg+LEE011 600mg: MEK162 45mg BID+LEE011 600mg QD
- Phase 2 - Dose Expansion Phase: The dose-expansion phase was initiated with a newly recruited group of patients.
  Binimetinib 45 mg BID + ribociclib 200 mg QD on 28-day schedule
Arm/Group | Phase 1b - 28 Day MEK162 45mg+LEE011 200mg | Phase 1b - 28 Day MEK162 45mg+LEE011 250mg | Phase 1b - 28 Day MEK162 30mg+LEE011 300mg | Phase 1b - 28 Day MEK162 45mg+LEE011 300mg | Phase 1b - 21 Day MEK162 30mg+LEE011 200mg | Phase 1b - 21 Day MEK162 45mg+LEE011 200mg | Phase 1b - 21 Day MEK162 30mg+LEE011 300mg | Phase 1b - 21 Day MEK162 45mg+LEE011 300mg | Phase 1b - 21 Day MEK162 45mg+LEE011 450mg | Phase 1b - 21 Day MEK162 45mg+LEE011 600mg | Phase 2 - Dose Expansion Phase
All-Cause Mortality (participants affected / at risk) | 3/16 | 0/3 | 1/4 | 1/6 | 0/5 | 1/6 | 0/2 | 0/4 | 0/9 | 1/6 | 23/41
Serious Adverse Events (participants affected / at risk) | 8/16 | 2/3 | 2/4 | 4/6 | 2/5 | 3/6 | 1/2 | 3/4 | 3/9 | 2/6 | 22/41
Other Adverse Events (participants affected / at risk) | 16/16 | 3/3 | 4/4 | 6/6 | 5/5 | 6/6 | 2/2 | 4/4 | 9/9 | 6/6 | 41/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b - 28 Day MEK162 45mg+LEE011 200mg (N=16) | Phase 1b - 28 Day MEK162 45mg+LEE011 250mg (N=3) | Phase 1b - 28 Day MEK162 30mg+LEE011 300mg (N=4) | Phase 1b - 28 Day MEK162 45mg+LEE011 300mg (N=6) | Phase 1b - 21 Day MEK162 30mg+LEE011 200mg (N=5) | Phase 1b - 21 Day MEK162 45mg+LEE011 200mg (N=6) | Phase 1b - 21 Day MEK162 30mg+LEE011 300mg (N=2) | Phase 1b - 21 Day MEK162 45mg+LEE011 300mg (N=4) | Phase 1b - 21 Day MEK162 45mg+LEE011 450mg (N=9) | Phase 1b - 21 Day MEK162 45mg+LEE011 600mg (N=6) | Phase 2 - Dose Expansion Phase (N=41)
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 4
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood creatine phosphokinase (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chronic obstructive pulmonary (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Obstructive airways (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Slow speech (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hemiplegia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Retinal detachment (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rectal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Subileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chills (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Micturition frequency (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 2
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b - 28 Day MEK162 45mg+LEE011 200mg (N=16) | Phase 1b - 28 Day MEK162 45mg+LEE011 250mg (N=3) | Phase 1b - 28 Day MEK162 30mg+LEE011 300mg (N=4) | Phase 1b - 28 Day MEK162 45mg+LEE011 300mg (N=6) | Phase 1b - 21 Day MEK162 30mg+LEE011 200mg (N=5) | Phase 1b - 21 Day MEK162 45mg+LEE011 200mg (N=6) | Phase 1b - 21 Day MEK162 30mg+LEE011 300mg (N=2) | Phase 1b - 21 Day MEK162 45mg+LEE011 300mg (N=4) | Phase 1b - 21 Day MEK162 45mg+LEE011 450mg (N=9) | Phase 1b - 21 Day MEK162 45mg+LEE011 600mg (N=6) | Phase 2 - Dose Expansion Phase (N=41)
Oedema peripheral (General disorders) | 7 | 2 | 2 | 3 | 1 | 2 | 0 | 2 | 2 | 0 | 18
Fatigue (General disorders) | 6 | 1 | 3 | 0 | 3 | 5 | 2 | 1 | 3 | 2 | 15
Pyrexia (General disorders) | 2 | 2 | 1 | 0 | 2 | 1 | 0 | 2 | 2 | 2 | 11
Chills (General disorders) | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 6
Aeaemia (Blood and lymphatic system disorders) | 5 | 2 | 2 | 4 | 2 | 1 | 0 | 1 | 4 | 0 | 10
Neutropenia (Blood and lymphatic system disorders) | 3 | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 4 | 3 | 5
Nausea (Gastrointestinal disorders) | 6 | 2 | 3 | 4 | 4 | 3 | 2 | 1 | 1 | 1 | 22
Diarrhoea (Gastrointestinal disorders) | 6 | 2 | 2 | 4 | 3 | 4 | 2 | 2 | 3 | 5 | 21
Vomiting (Gastrointestinal disorders) | 4 | 3 | 4 | 3 | 3 | 2 | 1 | 1 | 2 | 2 | 14
Constipation (Gastrointestinal disorders) | 3 | 1 | 2 | 3 | 0 | 1 | 0 | 1 | 3 | 0 | 8
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 2 | 5
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1 | 2 | 1 | 1 | 3 | 0 | 4
Stomatitis (Gastrointestinal disorders) | 4 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 4
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 3
Leukopenia (Blood and lymphatic system disorders) | 4 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 3 | 1 | 3
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 2 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Granulocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cardio-respiratiory arrest (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chorioretinopathy (Eye disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Retinal detachment (Eye disorders) | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 6
Vision blurred (Eye disorders) | 2 | 0 | 2 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 0
Retinopathy (Eye disorders) | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 0
Macular oedema (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 5
Subretinal fluid (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 5
Dry eye (Eye disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Detachment of retinal pigment epithelium (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Chorioretinal disorder (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Periorbital oedema (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Retinal disorder (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 2 | 2 | 0 | 1 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Face oedema (General disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Pain (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Astenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of the sponsor's agreements with its investigators may vary. However, the sponsor does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e., data from all sites) in the clinical trials.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-05-16): https://cdn.clinicaltrials.gov/large-docs/72/NCT01781572/SAP_000.pdf
  • Study Protocol (2015-08-26): https://cdn.clinicaltrials.gov/large-docs/72/NCT01781572/Prot_001.pdf